CLINICAL TRIAL: NCT03796611
Title: Phenotypic and Functional Study of 4BL B Cells in Multiple Sclerosis (MS)
Acronym: 4BLMS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_04; 2017-A00835-48 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Multiple Sclerosis
Keywords: immunology; B cells
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sampling and Cerebrospinal fluid at baseline and five sequential blood sampling for MS groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- multiple sclerosis patient: MS is defined according to McDonald criteria 2017. MS patients included have a disease duration of less than 1 year
- other neurological inflammatory disease: autoimmune encephalitis, myasthenia gravis, chronic inflammatory demyelinating polyradiculitis
- neurological non inflammatory disease: benign intracranial hypertension, degenerative disorder
- healthy controls: transfusion volunteers from transfusion center

SUMMARY:
Recent works highlight the B cells involvement in multiple sclerosis (MS) pathology but their role remains poorly understood. It was previously described that activated memory B cells called 4BL due to the increased expression of 4-1BBL, an activation marker, induce pro-inflammatory response by activating T CD8+ lymphocytes. Those 4BL cells are also described in systemic inflammation in 80 years old people explaining the poor efficiency of vaccination in that sub population. Those 4BL cells can also induce anti-tumoral T cell response.

The hypothesize is that 4BL may induce a pathogenic inflammatory response in MS.

DETAILED DESCRIPTION:
the aim to compare the proportion of peripheral (blood) 4 BL cells but also 4-BL cells in cerebro spinal fluid (CSF) in MS compared to healthy controls and to other inflammatory neurological disease but also non inflammatory neurological disease.

For all groups of patients and controls it will collect blood and CSF only once (at diagnosis time for patients).

Blood collect from healthy controls will come from transfusion volunteers and we won't have CSF from them.

For patients from the MS group, the blood collect will be sequential at diagnosis, 3, 6, 12 and 24 months after during the follow up.

In the blood and CSF we will evaluate:

* percentage of 4 BL cells. 4 BL cells are found using cytometric parameters
* capacity of 4 BL cells to induce inflammatory response in vitro: percentage of induced activated TCD8 proliferation after cell culture using extracellular and intracellular cytometric parameters

ELIGIBILITY:
Inclusion Criteria for MS group:

* MS defined by McDonald 2017 criteria with a disease duration of less than 1 year
* between 18 and 60 years old patients
* naïve of any immune therapy or steroid intake
* patients who signed consent to the study

Inclusion Criteria for controls with inflammatory of non inflammatory neurological disease:

* patients who signed consent to the study
* between 18 and 60 years old patients
* naïve of any steroid intake or immune therapy

Inclusion criteria for healthy controls:

* control who signed consent at transfusion center for their blood collect to be used for study
* between 18 and 60 years old patients
* naïve of any steroid intake or immune therapy

Exclusion Criteria:

* pregnancy or breast-feeding
* patients or controls unable to sign the consent or to consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: MS patients and controls: healthy controls and patients having non-MS neurological inflammatory disease and patients having other non inflammatory neurological disease.
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
the percentage of 4 BL cells in blood between MS patients and healthy controls | Baseline: one session
  4 BL are defined using cytometric parameters

SECONDARY OUTCOMES:
the percentage of 4 BL cells in blood between MS patients and patients with inflammatory and non inflammatory neurological disease | Baseline: one session
  4 BL are defined using cytometric parameters
the percentage of 4 BL cells in CSF between MS patients and patients with inflammatory and non inflammatory neurological disease | Baseline: one session
  4 BL are defined using cytometric parameters
to analyse over time the evolution of 4BL percentages in blood in MS patients | 5 blood collection at baseline, 3, 6, 12, and 24 months after baseline
  4 BL are defined using cytometric parameters

OTHER OUTCOMES:
biological bank with mononuclear cells from all the groups fo that study | through study completion, an average of 2 years
  to constitute at Baseline a biological bank with mononuclear cells from all the groups fo that study

CONTACTS AND LOCATIONS:
Overall Officials: Hélène ZEPHIR, MD, PhD, Principal Investigator — University Hospital, Lille